CLINICAL TRIAL: NCT04547777
Title: A Phase 1 Trial of D2C7-IT in Combination With an Fc-engineered Anti-CD40 Monoclonal Antibody (2141-V11) Administered Intratumorally Via Convection-Enhanced Delivery Followed by Perilymphatic Injections of 2141-V11 and Assessment of the Tumor Monorail for Adult Patients With Recurrent Malignant Glioma
Brief Title: Phase 1 Trial of D2C7-IT in Combination With 2141-V11 for Recurrent Malignant Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Darell Bigner (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor-Investigator, Darell Bigner, E. L. and Lucille F. Jones Cancer Distinguished Research Professor, in the School of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00104852
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Glioma, Malignant
Keywords: D2C7; D2C7-IT; Glioblastoma; Glioma; 2141-V11; Pro00104852; Duke; Rockefeller; CD40; epidermal growth factor receptor (EGFR); EGFR; Landi
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — D2C7-(scdsFv)-PE38KDEL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- D2C7-IT + 2141-V11 (Experimental): Single D2C7-IT intratumoral infusion (4613.2 ng/mL in 36 mL) over 72 hours followed by single 2141-V11 (3.0 mg, RP2D established prior to V5.0) infusion (5 dose levels) over 7 hours. This will be followed 2 weeks later by initiation of CPL subcutaneous injections of 2141-V11 at 2.0 mg, which will be repeated again 2 weeks later and then every 3 weeks for 1 year.
  Interventions: Drug: D2C7-IT; Drug: 2141-V11
- D2C7-IT + 2141-V11 and Tumor Monorail Device (TMD) Placement (Experimental): Patients who meet eligibility and agree with TMD placement will have the TMD implanted approximately 14 days prior to D2C7-IT infusion. Intraoperative CT will be performed post implant to ensure device location accuracy and check for hemorrhage. Prior to catheter insertion for D2C7-IT infusion, the first tumor/fluid sampling through the TMD will occur. Repeated tumor/fluid sampling via the TMD will occur prior to every 2141-V11 perilymphatic infusion, i.e., approximately 2 weeks (+ 1 week) after D2C7-IT and then every 3 weeks for 1 year.
  Interventions: Drug: D2C7-IT; Drug: 2141-V11

INTERVENTIONS:
Drug: D2C7-IT — D2C7-IT intratumoral infusion
Drug: 2141-V11 — 2141-11 intratumoral infusion
  Other Names: anti-CD40

SUMMARY:
This is a phase 1 study of an anti-CD40 monoclonal antibody (2141-V11) in combination with D2C7-IT for patients with recurrent World Health Organization (WHO) grade III or IV malignant glioma at the Preston Robert Tisch Brain Tumor Center (PRTBTC) at Duke.

DETAILED DESCRIPTION:
Within this study, a maximum of 30 patients with recurrent WHO grade III and IV malignant glioma will receive D2C7-IT and 2141-V11 to determine the impact of the combination of D2C7-IT and 2141-V11 on safety. D2C7-IT and 2141-V11 will be delivered sequentially directly into the tumor by Convection Enhanced Delivery (CED) using an intracerebral catheter placed within the enhancing portion of the tumor. Based on phase 1 studies of D2C7-IT alone and D2C7-IT in combination with atezolizumab in adult patients with recurrent glioblastoma (GBM), the amount of D2C7-IT to be delivered will be 4613.2 ng/mL (36 mL). 2141-V11 will be dose escalated during the study to determine the maximum tolerated dose (MTD) when used in combination with D2C7-IT.

Upon approval of v.9.0 of the protocol, patients will be eligible to receive D2C7-IT + 2141-V11 (via CED and CPL) with or without prior implantation of Tumor Monorail Device (TMD). Patients will be stratified into the following subgroups:

* Subgroup #1: Patients accrued before Protocol Version v.5.0
* Subgroup #2: Patients accrued after Protocol Version v.5.0 who did not have a TMD implanted.
* Subgroup #3: Patients accrued after Protocol Version v.9.0 for whom a TMD implantation was initiated.

Patients who enroll in subgroup #3, once identified as safe to proceed with the TMD (e.g. smaller tumor) and after obtaining their agreement, will receive the TMD approximately 14 days before intracranial D2C7-IT + 2141-V11 infusion in a modified 3+3 design (a minimum of 3 patients and a maximum of 9). All patients who do not meet inclusion criteria for the TMD and/or refuse to receive the TMD, will be treated under subgroup #2 and will proceed directly to CED catheter implantation followed by D2C7-IT + 2141-V11.

For patients enrolled subgroup #3, an initial 3 patients will be observed for safety before enrolling the next cohort of 3 patients. Intraoperative CT will be performed post implant to ensure device location accuracy and to check for hemorrhage. Prior to CED catheter insertion for D2C7-IT + 2141-V11 infusion, the first tumor/fluid sampling through the TMD will occur. Repeated tumor/fluid sampling via the TMD will occur before every perilymphatic injection of 2141-V11, i.e., approximately 2 weeks (+ 1 week) after D2C7-IT, which will be repeated again 2 weeks later and then every 3 weeks for 1 year. If fewer than 2 of the first 3 patients who receive the TMD experience an unacceptable adverse event within 14 days of TMD implantation, 3 more patients will receive the TMD. The TMD sampling time can be adjusted from every 3 weeks to every 6 weeks (i.e., every other 2141-V11 infusion) if not enough cellular and genomic material is sampled in the first cohort. With protocol version 10.0, patients who have completed 1 year of CPL subcutaneous injections of 2141-V11 at 2.0 mg every 3 weeks, who benefit from the therapy, and desire to continue on therapy will receive CPL subcutaneous injections of 2141-V11 at 2.0 mg every 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Study population:

   1. Subgroup #2: Histopathologically confirmed recurrent supratentorial WHO grade 3 or 4 malignant glioma (high grade glioma with molecular features of glioblastoma will be eligible under WHO grade 4 malignant glioma)
   2. Subgroup #3: Histopathologically confirmed recurrent supratentorial WHO grade 4 malignant glioma (high grade glioma with molecular features of glioblastoma will be eligible under WHO grade 4 malignant glioma) and found amenable for Tumor Monorail Device (TMD) implantation as per the treating neurosurgeon
2. Patient or partner(s) meets one of the following criteria:

   1. Non-childbearing potential (i.e.) not sexually active, physiologically incapable of becoming pregnant, including people who are post-menopausal or surgically sterile. Surgically sterile people are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation or have had a vasectomy. Postmenopausal for purposes of this study is defined as 1 year without menses.; or
   2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g. a condom or diaphragm) used with spermicide.
3. Age ≥ 18 years of age at the time of entry into the study
4. Karnofsky Performance Score (KPS) ≥ 70%
5. Hemoglobin ≥ 9 g/dl prior to biopsy
6. Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion
7. Neutrophil count ≥ 1000 prior to biopsy
8. Creatinine ≤ 1.5 x normal range prior to biopsy
9. Total bilirubin ≤ 1.5 x ULN prior to biopsy (Exception: Participant has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
10. AST/ALT ≤ 2.5 x ULN
11. Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anticoagulation will be held in the perioperative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to biopsy.
12. At the time of biopsy, prior to administration of D2C7-IT, the presence of recurrent tumor must be confirmed by histopathological analysis
13. A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study
14. Able to undergo brain MRI with and without contrast

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding/chestfeeding
2. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
3. Patients with severe, active co-morbidity, defined as follow:

   1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
   3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
   4. Patients with known lung (forced expiratory volume in the first second of expiration (FEV1) < 50%) disease or uncontrolled diabetes mellitus
   5. Patients with albumin allergy
4. Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks), or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy
5. Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy
6. Patients may not have received treatment with tumor treating fields (e.g., Optune) ≤ 1 week prior to starting the study drug
7. Patients may not be less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation
8. Patients who have not completed all standard of care treatments, including surgical procedure and radiation therapy (Please note: For patients under 65 years old, standard radiation therapy is typically at least 59 Gy in 30 fractions over 6 weeks. For patients 65 years or older, standard RT is often reduced to a minimum 40 Gy in 15 fractions over 3 weeks.)

   1. If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial
   2. If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter methylation status is unknown at time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial
9. Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of active (growing) disease (active multifocal disease); extensive subependymal disease (tumor touching subependymal space is allowed); tumor crossing the midline or leptomeningeal disease
10. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the D2C7-IT infusion
11. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
12. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
13. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months
14. Only for patients in Subgroup #3 (TMD subgroup): Patients with known allergies to silicone, polyurethane and titanium, which are materials contained in the TMD

Subject Eligibility Salvage Treatment (Effective with Protocol Version v.5.0)

Before being allowed to proceed with salvage treatment, the subject must satisfy the following inclusion and exclusion criteria. This option is available only for patients treated prior to Protocol Version v.5.0 - Subgroup #1:

Inclusion Criteria Salvage Treatment

1. Patients must have a recurrence of their supratentorial WHO grade IV4 malignant glioma based on imaging studies with measurable disease requiring therapy other than per protocol allowed reduced dose bevacizumab
2. Patients must be ≥ 4 months since their intratumoral administration of D2C7-IT + 2141-V11
3. A new signed informed consent form for the treatment with 2141-V11 in the CPL area ipsilateral to the tumor approved by the Institutional Review Board (IRB) of record will be required. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of the injection of 2141-V11 in the CPL subcutaneous area.
4. If the subject is able to produce sperm and is sexually active, they are eligible to enter and receive treatment with 2141-V11 injected in the CPL subcutaneous area if their partner(s) meets the criteria outlined in sub-bullet a. below or if they or their partner(s) are using one of the methods of birth control outlined in sub-bullet b. below. If the subject is potentially able to become pregnant, they are eligible to enter and participate in this study if they meet the following criteria:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including people who are postmenopausal or surgically sterile). Surgically sterile people are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study, is defined as 1 year without menses); or
   2. Childbearing potential, has a negative serum pregnancy test at screening, and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g., birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g., a condom or diaphragm) used with spermicide.
   3. Please note: If the patient has had a vasectomy or is using a condom with spermicide, their partner does not need to use additional birth control noted in 4a and 4b.
5. Total bilirubin ≤ 1.5 x ULN prior to CPL injection (Exception: Participant has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
6. AST/ALT ≤ 2.5 x ULN prior to CPL injection.
7. Neutrophil count ≥ 1000 prior to CPL injection.
8. Platelet count ≥ 50,000/µL unsupported is necessary prior to CPL injection.
9. Creatinine ≤ 1.2 x normal range prior to CPL injection.

Exclusion Criteria Salvage Treatment

1. Patients who are pregnant or breastfeeding/chestfeeding
2. Patients with severe, active co-morbidity, defined as follow:

   1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
   3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
   4. Patients with known lung (forced expiratory volume in the first second of expiration [FEV1] < 50%) disease or uncontrolled diabetes mellitus
3. Karnofsky Performance Score < 60%
4. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the 2141-V11 injection in the CPL area
5. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with dose-limiting toxicity (DLT) within each dose level | 28 days after catheter removal
  DLTs are defined as any of the following events that are at least possibly, probably, or definitely attributable to study treatment (2141-V11 or the combination of D2C7-IT and 2141-V11) during dose escalation. As the optimal dose of D2C7-IT in monotherapy has been well established, only toxicity starting or increasing in grade at any time after the start of 2141-V11 will be considered for DLT definition.
Proportion of patients with unacceptable toxicity resulting from injections of 2141-V11 in the CPL area ipsilateral to the tumor | 28 days after catheter removal
  For the purpose of monitoring adverse events occurring with perilymphatic injections of 2141-V11, we will define an unacceptable toxicity as any adverse event that satisfies the definition of DLT.
The proportion of patients with Tumor Monorail Device (TMD)-related unacceptable adverse event | 14 days following TMD placement
  Unacceptable adverse events following TMD placement are defined as follows
  * Cerebral edema (grade 3 or higher) due to device implantation
  * New neurological symptoms (grade 3 or higher) that do not resolve within 2 weeks and not due to tumor progression
  * Device-related infection (grade 3 or higher)
  * Intracranial hemorrhage (grade 3 or higher)
  * Tumor mis-migration (extracranial extension)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD,FRCPC, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker S, McDowall C, Sanchez-Perez L, Osorio C, Duncker PC, Briley A, Swartz AM, Herndon JE 2nd, Yu YA, McLendon RE, Tedder TF, Desjardins A, Ashley DM, Gunn MD, Enterline DS, Knorr DA, Pastan IH, Nair SK, Bigner DD, Chandramohan V. Immunotoxin-alphaCD40 therapy activates innate and adaptive immunity and generates a durable antitumor response in glioblastoma models. Sci Transl Med. 2023 Feb 8;15(682):eabn5649. doi: 10.1126/scitranslmed.abn5649. Epub 2023 Feb 8. PMID 36753564
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials